CLINICAL TRIAL: NCT02166723
Title: Treatment of Long Persistent Atrial Fibrillation by Single Cryoballoon Ablation of the Pulmonary Veins, Left Atrial Roof Line and Ablation of Left Lateral Ridge From Within the Appendage
Brief Title: Persistent Atrial Fibrillation Cryoballoon Ablation
Acronym: PAFCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Estelle Torbey, MD, Staten Island University Hospital
Other Study IDs: SIUH13-007
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; Cryoballoon ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CRYOABLATION: Cryoballoon ablation will be applied to all patients with persistent atrial fibrillation. It consists on applying the Arctic Front Cryoballoon to the pulmonary veins and freezing the antrum. In addition debulking of the atrial roof will be performed by a single application of the cryoballoon to the left and right roof, the septal wall and the lateral ridge wall.
  Interventions: Device: Cryoballoon Ablation

INTERVENTIONS:
Device: Cryoballoon Ablation — . The goal was to isolate all 4 veins with application of cryoballoon on the ostium of the vein. A 28 mm balloon was used with centrifugal cooling system. The maximum temperature reached was between -45 C and -60 C to optimize irreversible isolation without causing extracardiac complications. A circular catheter (Achieve) was used to map electrograms in conjunction with the NavX ENSITE 3000, St Judes . Intracardiac ultrasound was used to measure the pulmonary vein diameter, check for intraoperative complications, determine complete occlusion of the vein by the balloon and guide transeptal puncture. . In each patient the left atrium was debulked by applying cryoballoon
  Other Names: Arctic Front cryoballoon
Device: cryoballoon ablation — A 28 mm balloon was used with centrifugal cooling system. The maximum temperature reached was between -45 C and -60 C to optimize irreversible isolation without causing extracardiac complications. A circular catheter (Achieve) was used to map electrograms in conjunction with the NavX ENSITE 3000, St Judes . Intracardiac ultrasound was used to measure the pulmonary vein diameter, check for intraoperative complications, determine complete occlusion of the vein by the balloon and guide transeptal puncture. In each patient the left atrium was debulked by applying cryoballoon to the left and right sides of the left atrial roof and cryoablation of the left lateral ridge from within the left atrial appendage.
  Other Names: Arctic Front cryoballoon

SUMMARY:
Patients with persistent irregular heartbeats also called persistent atrial fibrillation usually have a lower probability of curing their arrhythmia with ablation with heat called radiofrequency then those with paroxysmal atrial fibrillation, as previous studies have shown.

The emerging ablation with freeze(cryoablation) has not been studied for persistent atrial fibrillation but has been proven to be efficient in the paroxysmal type.

We hypothesized that persistent atrial fibrillation will have a freedom of recurrence rate of 70% after use of cryoablation at one year of follow up.

DETAILED DESCRIPTION:
This was a retrospective single center cohort study designed to assess the freedom from recurrence of atrial fibrillation in the sample of patients with long persistent atrial fibrillation.

All patients who underwent cryoballoon ablation for atrial fibrillation at Staten Island University Hospital in the period ranging from January 2010 to 2013 were included in the study.

Data was collected from the electronic medical record as well as from the physician's office records after Institutional Review Board approval of the protocol

.Data collected included demographics, comorbidities pertaining to diabetes, heart failure, coronary artery disease, stroke occurrence, medications including antiarrhythmics and anticoagulants, procedural details including time of procedure and of fluoroscopy, vein ostial size, number of veins isolated, time to first recurrence after blanking period, complications of procedure and mortality. All patient identifiers were kept in a password protected computer.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in the registry and who have symptomatic persistent atrial fibrillation presenting to the institution who favor ablation as first line therapy instead of antiarrhythmics
* All patients with symptomatic persistent atrial fibrillation who have failed antiarrhythmic therapy.

Exclusion Criteria:

* Patients refusing follow up by event monitor.
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with persistent atrial fibrillation who present to staten island university hospital. Those who are listed treatment by cryoballoon ablation at the discretion of the operating physician will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Time to Recurrence of atrial fibrillation | within 1 year after the procedure
  Recurrent atrial fibrillation is defined as re occurrence of atrial fibrillation in episode of more than 3 seconds as documented by device monitoring., loop recorder, implanted devices or event monitor. Only episodes that reoccur after the blanking period of 3 month post ablation are considered as recurrence.

SECONDARY OUTCOMES:
Procedural time | 1 year
  The procedure time will be plotted against the date the procedure is performed to assess the improvement in operator skill.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Kowalski, MD, Study Director — Staten Island University Hospital; Estelle Torbey, MD, Principal Investigator — Staten Island University Hospital; Soad Bekheit, MD, Study Chair — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, New York, New York, United States

REFERENCES:
- [Background] Andrade JG, Khairy P, Guerra PG, Deyell MW, Rivard L, Macle L, Thibault B, Talajic M, Roy D, Dubuc M. Efficacy and safety of cryoballoon ablation for atrial fibrillation: a systematic review of published studies. Heart Rhythm. 2011 Sep;8(9):1444-51. doi: 10.1016/j.hrthm.2011.03.050. Epub 2011 Mar 30. No abstract available. PMID 21457789
- [Background] Kowalski M, Grimes MM, Perez FJ, Kenigsberg DN, Koneru J, Kasirajan V, Wood MA, Ellenbogen KA. Histopathologic characterization of chronic radiofrequency ablation lesions for pulmonary vein isolation. J Am Coll Cardiol. 2012 Mar 6;59(10):930-8. doi: 10.1016/j.jacc.2011.09.076. PMID 22381429